CLINICAL TRIAL: NCT05644080
Title: 68Ga/177Lu-PSMA Theranostics in Recurrent Grade 3 and Grade 4 Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 412811
Record Dates: First submitted 2022-11-15; First posted 2022-12-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: Patients with recurrent grade 3 and grade 4 glioma will be recruited for treatment with 177Lu-PSMA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga/177Lu-PSMA theranostics in recurrent grade 3 and grade 4 glioma (Experimental): Patients demonstrating a high tumor uptake of 68Ga-PSMA on the diagnostic PET/MRI examination in the screening part of the study are eligible for a standard of 3 cycles, with a possible extension to maximum number of 6 cycles, of 177Lu-PSMA radionuclide therapy sessions. SPECT/CT will be performed after each cycle of treatment for dosimetry calculations, while 68Ga-PSMA PET/MRI, quality-of-life schemes and clinical examinations will be used to monitor therapeutic effects during the therapy cycles and up to 1.5 year after treatment initiation. The main endpoints of the study are progression-free survival and overall survival.
  Interventions: Radiation: 177Lu-PSMA I&T

INTERVENTIONS:
Radiation: 177Lu-PSMA I&T — Patients demonstrating a high tumor uptake of 68Ga-PSMA on the diagnostic PET/MRI examination in the screening part of the study are eligible for a standard of 3 cycles, with a possible extension to maximum number of 6 cycles, of 177Lu-PSMA radionuclide therapy sessions. SPECT/CT will be performed after each cycle of treatment for dosimetry calculations, while 68Ga-PSMA PET/MRI, quality-of-life schemes and clinical examinations will be used to monitor therapeutic effects during the therapy cycles and up to 1.5 year after treatment initiation. The main endpoints of the study are progression-free survival and overall survival.

SUMMARY:
This interventional, clinical pilot-study will initiate and evaluate 68Ga/177Lu-PSMA theranostics in Norway as treatment alternative for patients with recurrent grade 3 and grade 4 gliomas. The main goal is to improve existing diagnostic and therapeutic methods in glioma management, and introduce a novel, well-tolerated radionuclide treatment that possibly can increase the overall survival and quality of life for a patient group that today have very short expected survival and no standard recommended therapy.

DETAILED DESCRIPTION:
Patients demonstrating a high tumor uptake of 68Ga-PSMA on the diagnostic PET/MRI examination in the screening part of the study are eligible for a standard of 3 cycles, with a possible extension to maximum number of 6 cycles, of 177Lu-PSMA radionuclide therapy sessions. SPECT/CT will be performed after each cycle of treatment for dosimetry calculations, while 68Ga-PSMA PET/MRI, quality-of-life schemes and clinical examinations will be used to monitor therapeutic effects during the therapy cycles and up to 1.5 year after treatment initiation. The main endpoints of the study are progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* A previous diagnosis of histologically confirmed WHO grade 3 or grade 4 glioma
* Radiologically (MRI) confirmed tumor relapse/progression ≥ 12 weeks since completed radiotherapy or suspicion of recurrence where inclusion in the theranostic part of study could be indicated
* Must be ≥ 18 years old
* Written informed consent for study participation
* Negative pregnancy test no longer than 14 days prior to enrollment
* Life expectancy > 12 weeks
* Karnofsky performance status ≥ 70% (must be able to care for self after radionuclide therapy)
* High tumor uptake on diagnostic imaging with 68Ga -PSMA.
* Tumor not amendable for radiotherapy or surgery, and treating oncologist think that there are no other preferable systemic therapy options (e.g temozolomide, PCV or lomustine monotherapy).
* Women of childbearing potential (WOCBP) defined as fertile, following menarche and until becoming post-menopausal unless permanently sterile must use adequate contraception. Permanent sterilization methods include hysterectomy, bilateral salpingectomy or bilateral oophorectomy. Adequate contraception in the current study will be the following:

  o Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
  * Intravaginal
  * transdermal
  * Progestogen-only hormonal contraception associated with inhibition of ovulation:
  * oral
  * injectable
  * implantable
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system ( IUS)
  * bilateral tubal occlusion
  * vasectomised partner
  * sexual abstinence
* Patient accept not to receive any other tumor directed treatment before 8 weeks after each 177Lu-PSMA injection.

Exclusion Criteria:

* Estimated GFR < 30 mL/min
* Platelet count <75 x109 /L
* White blood cells ≤ 2.5 x 109/L
* Neutrophil count < 1.5 x109 /L
* Hb < 8.0 g/dL
* Albumin ≤ 25 g/L
* Uncontrollable symptomatic epilepsy refractory to standard medication
* Pacemakers or defibrillators not compatible with 3T MRI
* No ability to obtain informed consent (e.g. due to severe dysphasia or cognitive deficits).
* Breastfeeding
* Pregnancy
* Hypersensitivity to the active substance or to any of the excipients
* Urinary and fecal incontinence (patient cannot have diaper needs)
* Significant medical or psychiatric illness that, in the investigator's opinion, would compromise the patient's ability to tolerate this therapy
* If previous radiotherapy and/or radionuclide therapy have resulted in absorbed doses >=23 Gy to any of the kidneys, or >= 25 Gy to any of the parotids, an individual assessment will be made by the nuclear medicine physician and medical physicist if patient can be included to the therapy part of the study.
* Concurrent investigational drugs or experimental therapy must be stopped at least 4 weeks prior to study entry
* Unwilling to accept potential challenge with xerostomia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 6 months after end of therapy
  Type, frequency and severity of adverse events assessed with the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Evaluation of efficacy of 177Lu- PSMA | 6 months after commencement of therapy
  Progression free survival (6 months) determined from date of commencement of 177Lu-PSMA therapy
Evaluation of efficacy of 177Lu- PSMA | 1 year after commencement of therapy
  Overall survival (1 year) determined from date of commencement of 177Lu-PSMA therapy
Adverse events | Day 1 and 6 months after end of therapy
  Change in score in the modified RAI-6 questionnaire.

SECONDARY OUTCOMES:
Evaluate radiation dose to tumor and critical organs | 7 days after commencement of therapy
  Calculation of absorbed doses to the tumor and kidneys, parotid glands, sublingual glands, submandibular glands, lacrimal glands, liver, spleen and red marrow for each therapy cycle as well as accumulated doses for all therapy cycles.
Tumor response | 8 weeks
  Tumor responses as assessed by contrast enhanced MRI according to response assessment in neuro oncology (RANO) criteria (50) (Attachment 3) and volume measurements.
Nano score | 8 weeks
  Neurologic exam (nano score)
Health related quality of life | 8 weeks
  Health-related quality of life EQ-5D scores
Karnofsky performance status | 8 weeks
  Karnofsky performance status
PSMA uptake versus progression free survival | 8 weeks
  Correlate 68Ga-PSMA uptake (SUV) to overall and image-based progression free survival.
Pretherapeutic PSMA uptake versus accumulated doses | 8 weeks
  Evaluate the possible correlation between the pretherapeutic uptake of 68Ga -PSMA (SUV) in tumors and salivary glands to accumulated doses received from therapeutic 177Lu-PSMA.
Tumor-to-parotis ratio threshold for indication of 177Lu-PSMA therapy | 8 weeks
  Establish an appropriate indication for 177Lu-PSMA therapy by measuring tumor:parotis-ratios in 68Ga-PSMA PET scans.
Change in PSMA uptake during treatment period versus overall survival | 8 weeks
  Measure changes in uptake (SUV) of 68Ga-PSMA during the treatment period and correlate to overall survival in order to evaluate the role of post-therapeutic 68Ga-PSMA PET in monitoring disease.

CONTACTS AND LOCATIONS:
Overall Officials: Tora Solheim, MD/PhD, Principal Investigator — St. Olavs hospital/NTNU
Locations (1):
- St. Olavs hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McBriar JD, Shafiian N, Scharf S, Boockvar JA, Wernicke AG. Prostate-Specific Membrane Antigen Use in Glioma Management: Past, Present, and Future. Clin Nucl Med. 2024 Sep 1;49(9):806-816. doi: 10.1097/RLU.0000000000005365. Epub 2024 Jul 1. PMID 38968568